CLINICAL TRIAL: NCT02645448
Title: Glycemic Responses and of the Autonomic Cardiac Function in Diabetes Type-2 Women Post Resistance Exercise of Different Intensities
Brief Title: Glycemic Responses and of the Autonomic Cardiac Function in Diabetes Type-2 Women Post Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do vale do São Francisco (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, LOUMAÍRA CARVALHO DA CRUZ, Principal Investigator, Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: UFSaoFrancisco
Record Dates: First submitted 2015-12-12; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus; Autonomic Diseases
Keywords: Resistance Exercise; Diabetes Mellitus; Heart Rate Variability
MeSH Terms: conditions — Diabetes Mellitus; Autonomic Nervous System Diseases | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resistance Exercise Low intensity (Other): Day 1 (Control Session)
  Day 2 (Resistance Exercise)
  Day 3 (Duration of effect)
  Interventions: Other: Resistance Exercise
- Resistance Exercise High intensity (Other): Day 1 (Control Session)
  Day 2 (Resistance Exercise)
  Day 3 (Duration of effect)
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Resistance Exercise — Control Session
  Resistance exercise at different intensities (40%1RM or 80%1RM)
  Duration of effect

SUMMARY:
The aim of this study was to investigate and correlate the glucose responses and VFC 24 hours after resistance exercise (RE) sessions at different intensities in women with type 2 diabetes (DM-2). Twelve women with DM-2 were invited to perform by one week in randomized order, two weeks interventions with experimental sessions: Session Control (CONT) without conducting RE, RE session (40% or 80% of one maximum repetition - 1RM) on day 2 and day 3 was observed the effect of the length of RE session by 11h. After that, initiated the experimental sessions, where after each of the analysis of glucose 24h by continuous monitoring system of glucose was performed, considering breakfast, lunch, dinner and sleep, and analysis performed of the RR series by a period of 48h. During control sessions, the subjects were seated comfortably for 40min and RE sessions, 40%1RM and 80%1RM, were performed in medium circuit 3 sets with 16 and 8 replications and recovery range between 60 exercises and 90seg , respectively, and between the circuits 120sec. It was observed that the concentration of glucose in the period of 24h after the session has been reduced to 40% 1RM vs. CONT and 80%1RM. Hyperglycemia was prevalent in the period 34h of the sessions CONT and 80%1RM, respectively , being different from the session 40%1RM. In postprandial times, shorter hyperglycemia was found in the session to 40% 1RM vs. CONT and 80% 1RM after breakfast, lunch and dinner. At the time of sleep, less time in hyperglycemia was found between sessions of 40% 1RM vs. 80% 1RM. Significant correlations (p <0.01) were found between glucose 24h with cardiac autonomic RRi variables, HF, LF and reason LF:HF.

DETAILED DESCRIPTION:
This study was a randomized cross-by blocks in accordance with CONSORT (Schulz et al., 2010).

In total, 12 women with DM-2, between 48 and 60 years old participated in the study, where they were informed of risks, benefits and objectives of the study and signed a consent form Clarified (IC) previously approved by the Ethics Committee and Ethics in Research and Studies (CEDEP) of the Federal University of São Francisco Valley (UNIVASF), Petrolina - PE, Brazil (No. 0005/180814 CEDEP).

Of the participants, 11 were taking oral hypoglycemic medication (metformin [n = 7], Sulphonylurea [n = 1] Metformin in combination with sulfonylurea [n = 3]) and performed only dietary control.

Before the first visit to the UNIVASF Exercise Physiology Laboratory, the participants underwent a resting ECG examination, which could only be submitted to the test of a one maximum repetition (1RM) and meetings after report of normality certified by cardiologist.

On the first visit to the lab, participants responded history about health history, physical activity level and risk stratification. Subsequently were performed anthropometric measurements of waist circumference, abdomen and hip, as well as height and body mass for subsequent calculation of body mass index.

Two weeks before starting the intervention, participants underwent familiarization with the exercise protocol for three alternate days. After 48 hours was performed the 1RM test in the following exercises: bench press on the machine (pectoral and anterior deltoid muscle), extensor chair (quadriceps muscle), Flying (pectoral muscle), flexor chair (muscle biceps femoris, semitendinosus and semimembranosus), Pull High ahead (posterior muscles of the torso and biceps), leg press (quadriceps and gluteus), sitting Remada (posterior muscles of the torso and biceps) in equipment of Evidence® mark (Cachoerinha / RS - Brazil) and Physicus® (Auriflama / SP - Brazil).

After the 1RM test, participants received guidance in relation to food intake and the practice of daily physical activity, and that, 48 hours before the first day of intervention, do not ingest drinks contained alcohol and caffeine.

In the days of the sessions, participants fasted, they went to the lab, where they received a standard breakfast containing 285 kcal, 45g and (180 kcal) carbohydrate, 6 g (24 kcal) of protein and 9 g (81 kcal) of fat. Also they were asked to maintain the same diet during the two-week intervention and record consumption in a food diary, which was later analyzed and calculated by a trained nutritionist, using Microsoft Excel® software and the Brazilian Table of Food Composition.

It was also recommended that the main meals were taken at the same time of day (Breakfast between 7:00 and 7:20h; lunch between 12:00h and 14:00h and Dinner between 18:00h and 20:00h). The energy intake and consumption of daily macronutrients did not differ between sessions as shown in Table 2. During the days of intervention participants were instructed to refrain from any exercise and / or strenuous physical labor.

The glucose sensor (Sof-sensor, Medtronic Minimed, Inc., Northridge, CA, USA) has been installed the day before the first session being inserted following manufacturer's instructions SMGG Guardian real-time (Medtronic Minimed, Inc., Northridge CA, USA), which consists of a transmitter sensor inserted through a needle into the abdominal subcutaneous tissue using a device (Sen-Seter, Medtronic Minimed, Inc., Northridge, CA, USA) and a monitor for reading with wireless radio frequency sensor. This system has been validated in DM control studies and complications.

After the installation, there were appropriate calibration of the equipment following the manufacturer's recommendations. During the monitoring period, capillary glucose samples were collected using a glucose monitor (Accu-Check Performa, Roche Diagnostics, Mannheim, Germany) to calibrate the SMCG, being held four times every 24 hours monitoring by the researcher. Participants were blinded with regard to measurements of SMCG and capillary glucose during calibrations.

The glucose concentrations were analyzed on day 1 (24 hours analysis to observe the effect of the control section), Day 2 (24h analysis to observe the effect of Resistance Exercise - RE on different intensities) and day 3 (11h analysis of the duration of effect RE at different intensities).

To evaluate the autonomic modulation is adopted the frequency meter of Polar® RS800CX model (Electo Oy, Kempele, Finland) with proven validity and reproducibility (Essner et al, 2013; Jonckheer-SHEEHY et al, 2012.).

The investigated autonomic indicators were: 1) straight-time domain from absolute average records of RR intervals (RRi) and; 2) the frequency domain method for spectral analysis by Fast Fourier Transformer (low frequency - LF normalized units as a marker of sympathetic activity, high frequency - HF also with normalized units as a marker of vagal activity, and the LF:. HF as a marker of sympathovagal balance). All indexes are described by the European Society of Cardiology (TASK FORCE HEART Variability, 1996) and all Analyses were performed in Kubios HRV Analysis Software version 2.0 (Biosignal Laboratory, University of Kuopio, Finland).

All participants took part in a randomized experimental study, which consisted of two intervention periods, with each period consisted of three days where on day 1 a control session (CONT) was held, day 2 to RE session (40% 1RM or 80% 1RM), day 3 to check the duration of the effect of exercise. Each intervention aimed to assess the impact of a workout on glycemic control in standardized food and free living conditions.

Initially the participants arrived at the laboratory in fasting at 7: 00 and at that time was provided to them a standardized breakfast containing 285kcal, breakfast period was between 7: 00 - 7: 20h. After this period, the volunteers were instructed again on the subsequent power the sessions and even at that time, the frequency meter Polar RS800CX has been installed for reading RRi during and post-session, totaling 24 hours of Heart Rate Variability (HRV) measurements.

Each participant performed four sessions: CONT, ER 40% 1RM and ER 80% 1RM, and the RE sessions at different intensities randomized by blocks, in food standardization and abstention from other types of exercise, but free living conditions while using SMCG polar and frequency meter. In each session glycemic and autonomic responses were analyzed by a 24-hour period started at each session.

All sessions lasted 60 minutes, consisting of 20 minutes of a pre-intervention period (rest) and control session 40min (day1) and session RE (day 2), and were performed at the same time of day between 8:00 and 9:00. During all sessions the participants were already under the glucose monitoring and VFC. At the end of each session, participants were released to daily routine always under the use of SMCG and frequency meter.

The experimental sessions were distributed in two weeks, being held on the 1st of each week a control session and on day 2 an RE session (40% 1RM and 80% 1RM). On day 3 no intervention was only observed for a period of 11h monitoring, the possible duration of the ER effect in the preceding day.

Pre-intervention: Before any intervention, the participants remained seated in the laboratory for a period of 20 minutes in a quiet room without interference from noise and temperature between 23-24ºC (SOUZA et al, 2013.). During this period, every 5 minutes, the concentrations of glucose through the SMCG and RRi through the frequency meter were obtained.

Intervention: The intensities of RE have been established based on the classification of the American College Sport Medicine and American Diabetes Association for individuals with DM-2, and categorized the low intensity with 40% 1RM and high intensity exercise with 80% 1RM (Colberg et al., 2010). RE sessions 40% and 80% 1RM addition control section (no RE) lasted 40 minutes each. For RE sessions it was held three circuits with 7 exercise each, in the same sequence the 1RM test (the machine bench press, leg extension Chair, Flying, flexor chair, high Pull ahead, leg press, seated row). For RE session at 40% 1RM were performed 16 repetitions of each exercise with an interval of 60 seconds between them and 120 seconds between circuits. For RE session at 80% 1RM were performed 08 repetitions of each exercise with an interval of 90 seconds between them and 120 seconds between circuits. The duration repeat the exercise both 40% and 80% 1RM was 3 seconds, 1 second in the concentric phase and 2 seconds in the eccentric phase of the movement. In CONT sessions participants remained seated in a comfortable chair, being in the same room of the ER sessions.

Post-intervention: At the end of each session the participants were released to daily routine, being oriented to record daily food intake (day 1) and equalize the same consumption in the following days (days 2 and 3) during the two weeks of intervention. Also, avoid performing exercises of any nature and make use of the medication in the same way in periods of intervention.

Data were expressed as mean ± SD (standard deviation). Data normality was confirmed by the Shapiro-Wilk test. The glucose values were used to determine the average concentration of glucose and the prevalence of hyperglycemia (blood glucose concentrations exceeded 160 mg.dL-1) both in 24 and in the postprandial different times: breakfast (08: 00 - 12: 00), lunch (13:00h - 18:00h), dinner (19:00h - 23:00h) and sleep (23:00h - 06:00h). Analysis of variance one way (ANOVA) with repeated measures was performed to determine differences in experimental conditions (CONT x 40% x 80% 1RM). Post-hoc Tukey's pair for identification of differences was used as an 'F' mean was obtained. Pearson's linear correlation test was also adopted to investigate the association between glucose and HRV. Significance was set at p confidence level <0.05. All statistical calculations were performed using the STATISTICA software for Windows v. 6.0 (StatSoft, Inc.)

ELIGIBILITY:
Inclusion Criteria:

* Being female, diagnosed with type 2 diabetes (DM-2) and be clinically stable, and be aged between 40 and 60 years.

Exclusion Criteria:

* Make use of exogenous insulin
* Have morbid obesity (BMI> 40 kg / m2)
* Provide uncompensated glucose and abnormalities in the electrocardiogram (ECG) at rest with suggestion of cardiac ischemia from above or below unevenness in the ST segment> 2mm or reversal in T wave
* Presenting heart disease
* Proliferative diabetic retinopathy
* Severe autonomic neuropathy
* Any limb amputation
* Uncontrolled hypertension (systolic> 160 mmHg and / or diastolic BP> 100 mmHg)
* Diabetic nephropathy (albuminuria ≥ 14mg / L or> 30mg / 24h) chronic renal failure (SBD, 2014; ADA, 2014)
* Osteo-myo-articular problems that limited the exercises and being a smoker.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Concentration of glucose and hyperglycemia prevalence | 24 hours
  Acute bout of resistance exercise at 40% 1RM (low intensity) reduced glucose concentrations and the prevalence of hyperglycemia in 73.1 ± 37.7% and 68.4 ± 51.1% compared to the sessions CONT40% and resistance exercise 80% 1RM (high intensity) respectively in 24h from each session.

SECONDARY OUTCOMES:
Heart Rate Variability | 24 hours
  In this study there was no difference between sessions of resistance exercise, during 24 hours, in any of the HRV indicators in the field of time and frequency.
Correlation between heart rate variability and glucose 24 hours | 24 hours
  Negative correlations between glucose 24 to the RR intervals and the parasympathetic modulation indicator HF, and positive correlations with the sympathetic modulation indicator LF and sympathovagal balance.

CONTACTS AND LOCATIONS:
Overall Officials: Loumaíra Carvalho da Cruz, Principal Investigator — Universidade Federal do vale do São Francisco

IPD SHARING:
Plan to Share IPD: No